CLINICAL TRIAL: NCT02839213
Title: The Effect of Hyoscine Butylbromide on Shortening of First and Second Stages of Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Kamal Mohamed Zahran, Prof, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBL
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Labor
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Hyoscine Butyl bromide group) (Active Comparator): The women will be given Hyoscine Butyl bromide
  Interventions: Drug: Hyoscine Butyl bromide
- group B (Saline group) (Active Comparator): The women will be given saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Hyoscine Butyl bromide
  Arms: group A (Hyoscine Butyl bromide group)
Drug: Saline
  Arms: group B (Saline group)

SUMMARY:
The management of normal labor is both an art and a science. For decades, health providers have worked to manage labor actively and safely, with the goal of shortening the duration of painful labor. Reduction of Cesarean sections and other fetal and maternal complications is also an important aspect of labor management.

The safety of active management of labor has been demonstrated by several prospective randomized clinical trials. A shorter duration of labor from admission to delivery has also been consistently reported in numerous studies of women treated with the active management protocol.Hyoscine butylbromide belongs to the parasympatholytic group of drugs and is a semisynthetic derivative of scopolamine. It is an effective antispasmodic drug without the untoward side effects of atropine. Hyoscine butylbromide is a quaternary ammonium compound and has peripheral anticholinergic action, but no central action as it does not cross the blood-brain barrier. Hyoscine butylbromide acts primarily by blocking the transmission of neural impulses in the intraneural parasympathetic ganglia of abdominal organs, apparently inhibiting cholinergic transmission in the synapses of the abdominal and pelvic parasympathetic ganglia, thus relieving spasms in the smooth muscles of gastrointestinal, biliary, urinary tract, and female genital organs, especially the cervico-uterine plexus, thus aiding cervical dilatation.

Spasmolytic drugs are frequently employed in delivery rooms to overcome cervical spasms and thus reduce the duration of labor.

Hyoscine butyl bromide has been used to shorten the duration of labor in several hospitals in the world. The mechanism by which it acts in the context of labor has not yet been elucidated, and evidence of its efficacy has been largely anecdotal.

Major studies have been carried out to evaluate the effects of the injectable or suppository form of Hyoscine butyl bromide on cervical dilatation; a majority of these studies demonstrated the efficacy of Hyoscine butyl bromide in augmenting labor. However, a few studies showed no effect of Hyoscine Butyl bromide on accelerating labor. In addition, some studies also used oxytocin in active management of labor, which would certainly affect the duration of labor and increase bias in the results. The specific objectives of this study will be to assess whether Hyoscine butyl bromide is effective in hastening cervical effacement and dilatation, thus shortening the duration of the first and second stages of labor with or without labor augmentation. We also intended to determine whether the use of Hyoscine butyl bromide in the first and second stages of labor has any associated increases in complications, such as an increase in blood loss or the rate of cesarean deliveries.

ELIGIBILITY:
Inclusion Criteria:

* All 18 -40 years.
* Singleton pregnancies.
* Vertex presentation.
* Term (gestational age between 37-41 weeks + 6 days).
* Spontaneous labor with either intact membranes or spontaneous rupture of membranes for less than 12 hours.

Exclusion Criteria:

* Previous uterine scarring including previous cesarean section.
* Cephalopelvic disproportion.
* Malpresentation.
* Antepartum hemorrhage.
* Multiple pregnancy.
* Induced delivery.
* Any medical disease.
* Prolonged premature rupture of the membrane (more than 12 hours).
* Epidural analgesia or receive any analgesic like pethidine.
* Pervious cervical cerclage.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The time of first and second stages of labor | 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes